CLINICAL TRIAL: NCT04899674
Title: An Open-label, Two-period Fixed Sequence Trial to Evaluate the Effect of Multiple Doses of BI 1358894 on the Pharmacokinetics of Bupropion in Healthy Volunteers
Brief Title: A Study in Healthy Men and Women to Test Whether BI 1358894 Influences the Amount of Bupropion in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1402-0018; 2020-006052-40 (EudraCT Number)
Record Dates: First submitted 2021-05-21; First posted 2021-05-24 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Healthy
MeSH Terms: interventions — Bupropion; TRPC inhibitor BI 1358894

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bupropion alone (Reference (R)) then BI 1358894 + bupropion (Test (T)) (Experimental)
  Interventions: Drug: Elontril; Drug: BI 1358894

INTERVENTIONS:
Drug: Elontril — Tablet
  Other Names: Bupropion hydrochloride
Drug: BI 1358894 — Film coated tablet

SUMMARY:
The main objective of this trial is to investigate the relative bioavailability of a single dose of bupropion when given alone (Reference) compared with co-administration (Test) with BI 1358894 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation
* Male subjects, or female subjects who meet any of the following criteria from at least 30 days before the first administration of trial medication until 30 days after trial completion:

  * Sexually abstinent
  * Use of adequate contraception, e.g. any of the following methods plus condom: implants, injectables, intrauterine device
  * A vasectomised sexual partner (vasectomy at least 1 year prior to enrolment)
  * Surgically sterilised (including hysterectomy)
  * Postmenopausal, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with levels of follicle stimulating hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion Criteria:

* Any finding in the medical examination (including safety laboratory, BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-09-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. Studies in products where Boehringer Ingelheim is not the license holder;
  2. Studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. Studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a phase I, open-label, two-period fixed sequence trial to evaluate the effect of multiple doses of BI 1358894 on the pharmacokinetics of bupropion in healthy volunteers.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Bupropion Alone (Reference (R)) Then BI 1358894 + Bupropion (Test (T)): Reference (R): Participants were administered on Day 1 of Visit 2 (Period: Reference) orally a single dose of 150 milligram (mg) of bupropion sustained release (SR) tablet (Elontril®) under fed conditions with 240 milliliter (mL) of water.
  Test (T): From Day -14 to Day 5 of Visit 3 (Period: Test) participants were administered orally once daily 2 film coated tablets of 50 mg of BI 1358894 (total dosage 100 mg/day) under fed conditions with 240 mL of water. On the 15th day of BI 1358894 administration (i.e. Day 1 of Visit 3 (Period: Test)) a single dose of 150 mg of bupropion was co-administered.
  The single-dose administrations of bupropion in Periods Reference and Test were to be separated by an interval of 21 days.
Period: Reference
Arm/Group | Bupropion Alone (Reference (R)) Then BI 1358894 + Bupropion (Test (T))
Started | 18
Completed | 18
Not Completed | 0
Period: Test
Arm/Group | Bupropion Alone (Reference (R)) Then BI 1358894 + Bupropion (Test (T))
Started | 18
Treated With BI 1358894 | 18
Treated With BI 1358894I and Bupropion | 17
Completed | 17
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The TS included all subjects who were randomised and treated with at least 1 dose of trial drug.
Arm/Group | Bupropion Alone (Reference (R)) Then BI 1358894 + Bupropion (Test (T))
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.7 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of Bupropion in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of bupropion in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) is presented.
  Time Frame: Within 3 hours (h) before and 1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 7 h, 8 h, 10 h, 12 h, 24 h, 48 h, 72 h, 96 h, 120 h after bupropion administration for the arm "bupropion alone (Reference (R))".
  Within 0.5 hours (h) before and 1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 7 h, 8 h, 10 h, 12 h, 24 h, 48 h, 72 h, 96 h, 120 h after bupropion administration for the arm "BI 1358894 + bupropion (Test (T))".
Time Frame: Up to 120 hours (h) after administration of bupropion (for detailed timeframe please see description).
Population: Pharmacokinetic (PK) parameter analysis set (PKS): This set included all subjects in the treated set (TS) who provided at least 1 PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Least Squares Mean (Standard Error); unit: hours * nanomole/Liter
Groups:
- Bupropion Alone (Reference (R)): Reference (R): Participants were administered on Day 1 of Visit 2 (Period: Reference) orally a single dose of 150 milligram (mg) of bupropion sustained release (SR) tablet (Elontril®) under fed conditions with 240 milliliter (mL) of water.
- BI 1358894 + Bupropion (Test (T)): Test (T): Participants were administered from Day -14 to Day 5 of Visit 3 (Period: Test) orally once daily 2 film coated tablets of 50 mg of BI 1358894 (total dosage 100 mg/day) under fed conditions with 240 mL of water. On the 15th day of BI 1358894 administration (i.e. Day 1 of Visit 3 (Period: Test)) a single dose of 150 mg of bupropion was co-administered.
Arm/Group | Bupropion Alone (Reference (R)) | BI 1358894 + Bupropion (Test (T))
Number analyzed (Participants) | 16 | 14
hours * nanomole/Liter | 2953 (NA) — Adjusted geometric standard error = 1.102. | 2795 (NA) — Adjusted geometric standard error = 1.104.
Statistical Analysis 1: Comparison: Bupropion Alone (Reference (R)) vs BI 1358894 + Bupropion (Test (T)); The statistical model used for the analysis of the primary endpoints was an Analysis of Variance (ANOVA) model. The model included effects accounting for the following sources of variation: 'subjects' and 'treatment'. The effect 'subjects' was considered as random, whereas the effect 'treatment' was considered as fixed; Test type: Other; Ratio of gMeans [%] = 94.6, 90% CI 2-sided [86.3 to 103.8] — Ratio of Geometric Least Squares Means (gMeans) was calculated as (gMean of "BI 1358894 + bupropion")/(gMean of "bupropion alone"). Intra-individual geometric coefficient of variation (gCV [%])=13.9

2. Primary Outcome: Maximum Measured Concentration of Bupropion in Plasma (Cmax)
Description: Maximum measured concentration of bupropion in plasma (Cmax) is presented.
  Timeframe: Within 3 hours (h) before and 1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 7 h, 8 h, 10 h, 12 h, 24 h, 48 h, 72 h, 96 h, 120 h after bupropion administration for the arm "bupropion alone (Reference (R))".
  Within 0.5 hours (h) before and 1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 7 h, 8 h, 10 h, 12 h, 24 h, 48 h, 72 h, 96 h, 120 h after bupropion administration for the arm "BI 1358894 + bupropion (Test (T))".
Time Frame: Up to 120 hours (h) after administration of bupropion (for detailed timeframe please see description).
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomole/Liter
Arm/Group | Bupropion Alone (Reference (R)) | BI 1358894 + Bupropion (Test (T))
Number analyzed (Participants) | 16 | 14
nanomole/Liter | 262 (NA) — Adjusted geometric standard error = 1.089. | 237 (NA) — Adjusted geometric standard error = 1.096.
Statistical Analysis 1: Comparison: Bupropion Alone (Reference (R)) vs BI 1358894 + Bupropion (Test (T)); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of gMeans[%] = 90.7, 90% CI 2-sided [74.3 to 110.7] — Ratio of Geometric Least Squares Means (gMeans) was calculated as (gMean of "BI 1358894 + bupropion")/(gMean of "bupropion alone"). Intra-individual geometric coefficient of variation (gCV [%])=31.5

3. Secondary Outcome: Area Under the Concentration-time Curve of Bupropion in Plasma Over the Time Interval From 0 to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of bupropion in plasma over the time interval from 0 to infinity (AUC0-∞) is presented.
  Time Frame: Within 3 hours (h) before and 1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 7 h, 8 h, 10 h, 12 h, 24 h, 48 h, 72 h, 96 h, 120 h after bupropion administration for the arm "bupropion alone (Reference (R))".
  Within 0.5 hours (h) before and 1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 7 h, 8 h, 10 h, 12 h, 24 h, 48 h, 72 h, 96 h, 120 h after bupropion administration for the arm "BI 1358894 + bupropion (Test (T))".
Time Frame: Up to 120 hours (h) after administration of bupropion (for detailed timeframe please see description).
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: hours * nanomole/Liter
Arm/Group | Bupropion Alone (Reference (R)) | BI 1358894 + Bupropion (Test (T))
Number analyzed (Participants) | 16 | 14
hours * nanomole/Liter | 3003 (NA) — Adjusted geometric standard error = 1.101. | 2855 (NA) — Adjusted geometric standard error = 1.103.
Statistical Analysis 1: Comparison: Bupropion Alone (Reference (R)) vs BI 1358894 + Bupropion (Test (T)); The statistical model used for the analysis of the primary endpoints was an Analysis of Variance (ANOVA). The model included effects accounting for the following sources of variation: 'subjects' and 'treatment'. The effect 'subjects' was considered as random, whereas the effect 'treatment' was considered as fixed; Test type: Other; Ratio of gMeans [%] = 95.1, 90% CI 2-sided [86.7 to 104.3] — Ratio of Geometric Least Squares Means (gMeans) was calculated as (gMean of "BI 1358894 + bupropion")/(gMean of "bupropion alone"). Standard deviation is actually intra-individual geometric coefficient of variation (gCV [%])=13.9

ADVERSE EVENTS:
Time Frame: Bupropion (BP): From administration (ad.) of BP+5 days of residual effect period (REP), up to 5 days(d). BI 1358894 + Bupropion: From ad. of BP on Day 1 of Visit 3 + 5 days of REP, up to 5 d. "BI 1358894 (BI) alone: From ad. of BI until ad. of BP or until last ad. prior to BP ad. + 14 d" "BI alone (continued): and from ad. of BP + 5 d of REP until last ad. of BI + 14 d of REP, up to 28d.
Description: Treated set (TS): The TS included all subjects who were randomised and treated with at least 1 dose of trial drug.
Groups:
- Bupropion: Participants were administered on Day 1 of Visit 2 (Period: Reference) orally a single dose of 150 milligram (mg) of bupropion sustained release (SR) tablet (Elontril®) under fed conditions with 240 milliliter (mL) of water.
- BI 1358894: Participants were administered from Day -14 to Day 5 (included) of Visit 3 (Period: Test) orally once daily 2 film coated tablets of 50 mg of BI 1358894 (total dosage 100 mg/day) under fed conditions with 240 mL of water.
- BI 1358894 + Bupropion: Participants were administered from Day 1 to Day 5 of Visit 3 (Period: Test) orally once daily 2 film coated tablets of 50 mg of BI 1358894 (total dosage 100 mg/day) under fed conditions with 240 mL of water. On Day 1 participants were co-administered a single dose of 150 mg of bupropion sustained release (SR) tablet (Elontril®) under fed conditions with 240 mL of water.
Arm/Group | Bupropion | BI 1358894 | BI 1358894 + Bupropion
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 4/18 | 9/18 | 3/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bupropion (N=18) | BI 1358894 (N=18) | BI 1358894 + Bupropion (N=17)
Headache (Nervous system disorders) | 2 | 8 | 3
Dizziness (Nervous system disorders) | 0 | 5 | 0
Coordination abnormal (Nervous system disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 3 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Body temperature increased (Investigations) | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/74/NCT04899674/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-13): https://cdn.clinicaltrials.gov/large-docs/74/NCT04899674/SAP_001.pdf